CLINICAL TRIAL: NCT04237922
Title: Replication of the TRITON-TIMI Antiplatelet Trial in Healthcare Claims Data
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-TRITON-TIMI
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Antiplatelet
MeSH Terms: interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clopidogrel 75 mg: Reference group
  Interventions: Drug: Clopidogrel 75mg
- Prasugrel 10 mg: Exposure group
  Interventions: Drug: Prasugrel 10mg

INTERVENTIONS:
Drug: Prasugrel 10mg — Prasugrel 10mg dispensing claim is used as the exposure group
  Groups: Prasugrel 10 mg
Drug: Clopidogrel 75mg — Clopidogrel 75 mg dispensing claim is used as the reference group
  Groups: Clopidogrel 75 mg

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as is possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Please see: https://drive.google.com/drive/folders/1WD618wrywYjEaXzfLTcuK-VCcnb6b-gV for full code and algorithm definitions.

Market availability of prasugrel in the U.S. started on 2009-07-10.

* For Marketscan: 2009-07-10 to 2017-12-31 (end of data availability).
* For Optum: 2009-07-10 to 2019-03-31 (end of data availability).

Inclusion Criteria:

* 1. Acute coronary syndrome based on the disease diagnostic criteria with planned PCI (ACS definition; one of the following):

  * 1a. Moderate to high risk Unstable angina: A history of chest discomfort or ischemic symptoms of 10 min or longer at rest, 72 h or less before randomization, with persistent or transient ST-segment deviation 1 mm or higher in one or more electrocardiogram (ECG) leads without elevation of creatine kinase-MB (CK-MB) or troponin T or I but with a TIMI risk score 321 or greater
  * 1b. II. Moderate to high-risk NSTEMI. A history of chest discomfort or ischemic symptoms of 10 min or longer at rest, 72 h or less before randomization with no evidence of persistent ST-segment elevation. Subjects must also have CK-MB or troponin T or I greater than the upper limit of normal (ULN) and a TIMI risk score 3 or greater. If CK-MB or troponin is not available, total CK 2 times or greater ULN is acceptable
  * 1c. III. STEMI. A history of chest discomfort or ischemic symptoms of greater than 20 minutes duration at rest, within 14 days or less randomization with one of the following ECG features:

    1. ST-segment elevation 1 mm or higher in 2 or more contiguous ECG leads
    2. New or presumably new left bundle branch block
    3. ST-segment depression 1 mm or greater in 2 anterior precordial leads (V1 through V4) with clinical history and evidence suggestive of true posterior infarction"
* 2. Legal age (and >18 y) and competent mental condition to provide written informed consent
* 3. For women of childbearing potential only, test negative for pregnancy between ACS presentation and enrollment (based on a urine or serum pregnancy test) and agree to use a reliable method of birth control during the study

Exclusion Criteria:

* Cardiovascular exclusion criteria

  * 1. Cardiogenic shock at the time of randomization
  * 2. Refractory ventricular arrhythmias
  * 3. New York Heart Association class IV congestive heart failure
* Bleeding risk exclusion criteria

  * 4. Fibrin-specific fibrinolytic therapy less than 24 h before randomization
  * 5. Non-fibrin-specific fibrinolytic therapy less than 48 h before randomization
  * 6. Active internal bleeding or history of bleeding diathesis
  * 7. Clinical findings, in the judgment of the investigator, associated with an increased risk of bleeding
  * 8. Any of the following:

    1. History of hemorrhagic stroke
    2. Intracranial neoplasm, arteriovenous malformation, or aneurysm
    3. Ischemic stroke within 3 months prior to screening
  * 9. International normalized ratio known to be greater than 1.5 at the time of screening
  * 10. Platelet count of less than 100000/mm3 at the time of screening
  * 11. Anemia (hemoglobin b10 g/dL) at the time of screening
* Prior/concomitant therapy exclusion criteria

  * 12. One or more doses of a thienopyridine 5 d or less before PCI
  * 13. Oral anticoagulation or other antiplatelet therapy that cannot be safely discontinued for the duration of the study
  * 14. Daily treatment with nonsteroidal antiinflammatory drugs (NSAIDs) or cyclooxygenase-2 inhibitors (COX-2 inhibitors)
* General exclusion criteria

  * 15. Investigative site personnel directly affiliated with the study or immediate family
  * 16. Employed by Eli Lilly and Company; Ube Industries Limited, Daiichi Sankyo Co.; The TIMI Study Group; Quintiles
  * 17. Treatment within the last 30 d with an investigational drug or are presently enrolled in another drug or device study
  * 18. Previously completed or withdrawn from this study or any other study investigating prasugrel
  * 19. Women who are known to be pregnant, have given birth within the past 90 d, or are breast-feeding
  * 20. Concomitant medical illness that in the opinion of the investigator is associated with reduced survival
  * 21. Known severe hepatic dysfunction
  * 22. Any condition associated with poor treatment compliance including alcoholism, mental illness, or drug dependence
  * 23. Intolerance of or allergy to aspirin, tilopidine, or clopidogrel
  * 24. May be unable to cooperate with protocol requirements and follow-up procedures

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve a new user, parallel group, cohort study design comparing prasugrel 90mg to clopidogrel 75mg. The patients will be required to have continuous enrollment during the baseline period of 180 days before initiation of prasugrel 90mg or a comparator drug (cohort entry date). Follow-up for the outcome (3P-MACE), begins the day after drug initiation.
Sampling Method: Non-Probability Sample
Enrollment: 43864 (Actual)
Dates: Start 2019-09-22 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Relative hazard of 3-P MACE (composite outcome of Stroke, MI, and Mortality) | Through study completion (a median of 276-312 days)
  Relative hazard of 3-point major adverse cardiovascular events (MACE), i.e., non-fatal myocardial infarction, non-fatal stroke, or all-cause/CV mortality- Please refer to uploaded protocol for full definition due to size limitations.

SECONDARY OUTCOMES:
Relative hazard of Hospital admission for MI | Through study completion (a median of 276-312 days)
  Relative hazard of Hospital admission for MI - Please refer to uploaded protocol for full definition due to size limitations.
Relative hazard of Hospital admission for stroke | Through study completion (a median of 276-312 days)
  Relative hazard of Hospital admission for stroke - Please refer to uploaded protocol for full definition due to size limitations.
Relative hazard of All-cause mortality/CV mortality | Through study completion (a median of 276-312 days)
  Relative hazard of All-cause mortality/CV mortality- Please refer to uploaded protocol for full definition due to size limitations.

OTHER OUTCOMES:
Relative hazard of Major bleeding (Control outcome) | Through study completion (a median of 276-312 days)
  Relative hazard of Major bleeding (Control outcome) - Please refer to uploaded protocol for full definition due to size limitations.
Relative hazard of Pneumonia (Control outcome) | Through study completion (a median of 276-312 days)
  Relative hazard of Pneumonia (Control outcome) - Please refer to uploaded protocol for full definition due to size limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham And Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Franklin JM, Patorno E, Desai RJ, Glynn RJ, Martin D, Quinto K, Pawar A, Bessette LG, Lee H, Garry EM, Gautam N, Schneeweiss S. Emulating Randomized Clinical Trials With Nonrandomized Real-World Evidence Studies: First Results From the RCT DUPLICATE Initiative. Circulation. 2021 Mar 9;143(10):1002-1013. doi: 10.1161/CIRCULATIONAHA.120.051718. Epub 2020 Dec 17. PMID 33327727

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/22/NCT04237922/Prot_SAP_000.pdf